CLINICAL TRIAL: NCT01644916
Title: "Consultation Liaison and Integrated Care for COPD Patients With Psychiatric Co-Morbidity"
Acronym: COPD_HSRG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other); Singapore General Hospital (Other); Alexandra Hospital (Other); St Luke's Hospital, Singapore (Other); Changi General Hospital (Other)
Responsible Party: Principal Investigator, A/Prof Ng Tze Pin, Research Director, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: COPD_HSRG_2010
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Anxiety; Depression
Keywords: COPD; Integrated care; IPCL
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depression | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual control (Other): Usual control will be provided with usual standard management of COPD and psychiatric comorbidities.
  Interventions: Procedure: Usual control
- Integrated care (Other): Integrated care will be provided with integrated care management.
  Interventions: Procedure: Integrated care

INTERVENTIONS:
Procedure: Integrated care — Integrated care will be provided with management of multifaceted group including, nurse educators, doctors, case manager and psychologists.
  Other Names: IPCL
  Arms: Integrated care
Procedure: Usual control — Usual control group will be provided with usual standard procedures for management of COPD and psychiatric comorbidities.
  Arms: Usual control

SUMMARY:
Chronic obstructive pulmonary disease (COPD) stands out among chronic diseases with its high and rising prevalence and mortality, poor quality of life, high re-hospitalization rates and societal burden of care. Current therapeutic and management practices are generally met with limited success. Research in recent years have highlighted the high level of psychiatric co-morbidity in COPD patients, and the major prognostic significance of anxiety/depression in COPD outcomes such as re-hospitalization, smoking cessation, quality of life, and survival. This suggests that addressing psychiatric and psycho-social aspects of care prominent in COPD patients may have strongly positive impact on outcomes, but the available evidence of effectiveness is limited.

The primary aim of the proposed research is to evaluate the effectiveness of a holistic disease management paradigm of psychiatric liaison consultation (CL) that integrates psychiatric and respiratory care to improve outcomes for COPD patients. This integrated psychiatric consultation liaison (IPCL) management paradigm includes the routine screening and structured collaborative care of anxiety and major depressive symptoms and depressive/anxiety disorder in COPD patients. We postulate that the IPCL care paradigm would reduce mood symptoms, increase smoking quit rates, reduce symptom burden and functional disability, and improve quality of life, while reducing rehospitalization, emergency department (ED) and unscheduled physician visits. A secondary aim is to evaluate its cost effectiveness by concurrently collecting resource utilization data.

DETAILED DESCRIPTION:
Specific Aims

The aim of the proposed research is to evaluate the effectiveness of a holistic disease management paradigm of) that integrates psychiatric and respiratory care (Integrated Psychiatric Consultation Liaison, IPCL) that addresses the high level of psychiatric co-morbidity in COPD patients to improve COPD outcomes.

Methods

Patient population Inpatients and specialist outpatients with established clinical diagnosis of chronic obstructive pulmonary disease (COPD).

Settings

Hospital based specialist outpatient and inpatient acute care and step-down care facilities in four hospitals (NUHS, AH, SGH and CGH) and one community hospital (SLH).

The site PIs from each hospital are Lim Tow Keang (NUHS),Loo Chian Min (SGH),K. Narendran (CGH), Gerald Chua (AH) and Tan Boon Yeow (SLH).

Study design Parallel group, randomized, controlled trial.

Eligible individuals are randomly assigned (1:1 ratio) to either:

1. Integrated Psychiatric Consultation Liaison (IPCL) care (N=450);
2. Usual care. Patients in this group will receive usual standard care (N=450).

Baseline screening and assessment. Prior to randomization to either IPCL or UC arm, COPD patients are screened for anxiety /depression using the Hospital Anxiety and Depression Scale (HADS, see below for details).21.For patients with high HADS scores(≥8), a semi-structured diagnostic assessment will be immediately performed using Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I for DSM-IV22 by an advanced practice nurse (APN) and the provisional diagnosis of anxiety and/or major depressive disorder will be confirmed by a psychiatrist, Cases with significant anxiety or depressive symptomatology that do not meet DSM-IV threshold criteria are classified as subsyndromal cases.

Randomization. After informed consent is signed and patient eligibility is confirmed, the patient will be randomized in a 1:1 ratio to either the intervention arm receiving IPCL care or the control arm receiving usual care. Stratification by center is used to ensure balance between the two arms across centers. Random permuted blocks are used to ensure balance over time. The block length is determined by the study statistician. The patient will be assigned an individual number upon randomization. This assigned randomized number will identify the patient and will be used for all documentation for this patient in this study. The list of randomizations will go through Singapore Clinical Research Institute (SCRI). Randomization may be done via the following options: (i) Direct web randomization: Authorized study center personnel will randomize the patient via a password-protected internet web site available 24 hours a day; (ii) Envelope Randomization: In case of web downtime due to technical error, site personnel may randomize patients using the back-up envelopes that will be provided upon activation of the site.

IPCL Care Group For patients who are randomly allocated to the IPCL arm,

1. Routine active screening and diagnosis of psychiatric co-morbidity using HADS followed by appropriate SCID interview by a trained APN, and confirmation by a consultant psychiatrist, will be performed at 3 monthly intervals during unscheduled and scheduled outpatient consultation or follow up visits and at each hospital admission.
2. The appropriate management of psychiatric and psycho-social problems will be performed by a multi-disciplinary care team that includes the respiratory physician, psychiatrist, advanced practice nurse and nurse clinicians
3. The APN and nurse clinician perform critical roles as case manager and patient educator. Psychoeducation is a critical care process component that will aim to ensure that the majority (over 70%) of COPD patients in the IPCL group with psychological symptoms will accept psycho-social and psychiatric care, in contrast to a large majority of patients who will conventionally refuse care, particularly in the UC group.
4. The treatment of cases will accord with recommended treatment guidelines for anxiety/depression, and individualized for each patient according to a treatment plan drawn up by the psychiatrist, with the agreement of the respiratory physician. Treatment and care management of mild depressive symptomatology, psycho-social problems, or severe major depression and/or anxiety disorder will include appropriate pharmacologic and/or non-pharmacologic therapies (such as cognitive and/or behavioural therapy) and psycho-social support.
5. Where pharmacologic treatment is indicated, the preferred drugs are SSRI antidepressants prescribed according to local standard dosages. The recommended first line of treatment is Fluoxetine, a dose of 20 mg/day or Escitalopram (10 to 20 mg/day). Alternatively, patients who do not respond to Fluoxetine or Escitalopram after 4 weeks, or who have intolerable side effects may be prescribed Venlafaxine XR, 75/mg/day, increased to 150-225 mg/day OR Mirtazapine (15mg/day, increased to 30-45 mg/day). If no response, mood stabilizer or electro convulsive therapy (ECT) or psychosocial intervention will be added on with the medication (Figure 2).
6. Non-drug psychotherapy will be provided either by the psychiatrist or psychological counselor where appropriate (for most patients with only depressive or anxiety symptomatology).
7. The case manager will liaise with medical social worker for financial and other community services support.
8. The nurse educator will provide standard patient education and behavioural modification including information about disease and medications for both COPD and depression, and changing attitudes and behaviour particularly in regard to smoking cessation and medication adherence, and general psycho-social supportive counseling.
9. Appropriate existing and redesigned treatment algorithms and management protocols will be put together and provide a sourcebook for drawing up individual care plans.
10. Routine monitoring and outcomes assessments is integrated as part of IPCL care and performed at 3 or 6 monthly intervals as appropriate: these include perceived symptoms of breathlessness, exercise tolerance, spirometric measurement (12 month), smoking cessation, HADS, SGRQ quality of life, acute COPD exacerbations, rehospitalization(s), emergency department visits, and unscheduled physician visits etc.(see schedule).
11. Ad hoc follow up visits are scheduled at any appropriate times for therapeutic monitoring and responses.
12. The management of COPD will proceed as usual according to standard clinical practice for COPD.

Usual Care Control Group. For patients who are randomly allocated to the UC Control Group,

1. The presence of psychiatric co-morbidity will be identified under standard conditions by usual care team, with the appropriate psychiatric consultation-liaison referrals and treatment effected as deemed necessary.
2. Treatment and care management of psychiatric and psycho-social problems will include appropriate pharmacologic and/or non-pharmacologic therapies and psycho-social support, in accordance with standard recommended guidelines and practices for both COPD and anxiety/depression.
3. The assessment of trial outcomes performed at 3 or 6 monthly intervals as appropriate (perceived symptoms of breathlessness, exercise tolerance, spirometric measurement, smoking cessation, HADS, SGRQ quality of life, acute COPD exacerbations, rehospitalization(s), emergency department visits, and unscheduled physician visits etc.) is also performed, but is not an integral part of Usual Care.
4. Ad hoc outpatient follow up visits are scheduled at any appropriate times for therapeutic and other care monitoring and responses.
5. The management of COPD will proceed as usual according to standard clinical practice for COPD.

To mimic prevailing conditions of healthcare financing and delivery, payments for referrals to hospital psychiatrists for treatment, drugs and psychotherapy, regardless of allocation to IPCL or UC group, will be borne by the patients using existing avenues of health service financing (Medisave, Medishield, and/or out-of-pockets) as appropriate.

Trial related scheduled assessments of outcome measures All participants in both IPCL and UC control arms will be assessed at baseline, 3 months, 6 months, 9 months and 12 months for the following trial related outcomes. We define loss to follow-up (LTFU) as incomplete ascertainment of the primary outcome for subjects randomized in the trial. Operationally, LTFU is defined as absence from at least 2 consecutive assessments (>6 months).

Statistical Analysis

Primary effectiveness end-points

* HADS score
* Breathlessness (MRC Index)
* Six-minutes walking distance
* Borg's scale
* FEV1, FEV1/FVC, PEFR, SpO2
* BODE Index
* Smoking quit rates
* Functional health and quality of life (SGRQ scores, CAT score, quality-adjusted life years (QALY))
* Acute COPD exacerbations
* Emergency department visits
* Unscheduled physician visits
* Re-hospitalization(s)

Secondary effectiveness end points:

* Resource use and direct costs of care:
* 1. Resource use include inpatient service use (No. of times hospitalized and total days in hospital) , outpatient service use (physician visits consisting of GP visits and specialist visits,) and medication use( usage of any or specific drug classes)
* 2. Direct costs of care include costs for outpatient medical and mental health care, inpatient medical and mental health services and medication.
* Mortality
* COPD medication adherence
* Psychiatric medication adherence

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and specialist outpatients from: NUHS, SGH, CGH, SLH and AH.
* Clinical diagnosis of chronic obstructive pulmonary disease (COPD) based on history, physical examination, spirometry, measurement of arterial blood gases, and chest radiographs, that meets the criteria for COPD as defined in the Global Initiative for Chronic Obstructive Lung Disease (GOLD).
* COPD patients include cases of all grades of severity, and co-morbidity, without restriction.
* Participants provide written informed consent.

Exclusion Criteria:

* Known diagnosis of a psychiatric disorder that is under treatment.
* Terminally ill COPD patients who are unable to complete baseline assessments.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
HADS score | over 12 months
  Anxiety and depression symptoms and diagnosis

SECONDARY OUTCOMES:
Resource use and direct costs of care | over 12 months
  Resource use include inpatient service use (No. of times hospitalized and total days in hospital) , outpatient service use (physician visits consisting of GP visits and specialist visits,) and medication use( usage of any or specific drug classes)and costs for resource use over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ng T Pin, MD, Principal Investigator — National University of Singapore
Locations (1):
- National University Hospital System, Singapore, Singapore

REFERENCES:
- [Background] Ng TP, Niti M, Tan WC. Trends and ethnic differences in COPD hospitalization and mortality in Singapore. COPD. 2004 Apr;1(1):5-11. doi: 10.1081/COPD-120028702. PMID 16997734
- [Background] Niti M, Ng TP, Kua EH, Ho RC, Tan CH. Depression and chronic medical illnesses in Asian older adults: the role of subjective health and functional status. Int J Geriatr Psychiatry. 2007 Nov;22(11):1087-94. doi: 10.1002/gps.1789. PMID 17407107
- [Background] Ng TP, Niti M, Fones C, Yap KB, Tan WC. Co-morbid association of depression and COPD: a population-based study. Respir Med. 2009 Jun;103(6):895-901. doi: 10.1016/j.rmed.2008.12.010. Epub 2009 Jan 10. PMID 19136238
- [Background] Cao Z, Ong KC, Eng P, Tan WC, Ng TP. Frequent hospital readmissions for acute exacerbation of COPD and their associated factors. Respirology. 2006 Mar;11(2):188-95. doi: 10.1111/j.1440-1843.2006.00819.x. PMID 16548905
- [Background] Ng TP, Niti M, Tan WC, Cao Z, Ong KC, Eng P. Depressive symptoms and chronic obstructive pulmonary disease: effect on mortality, hospital readmission, symptom burden, functional status, and quality of life. Arch Intern Med. 2007 Jan 8;167(1):60-7. doi: 10.1001/archinte.167.1.60. PMID 17210879
- See also: department of psychological medicine, gerontological research programme — http://www.nus.edu.sg